CLINICAL TRIAL: NCT03966482
Title: Exercise Of Semi-Occluded Vocal Tract In Velopharyngeal Dysfunction In Patients With Cleft Palate : Effects Of Short-Term
Brief Title: Semi-occluded Vocal Tract Exercise in Velopharyngeal Dysfunction in Patients With Cleft Palate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49953815.4.0000.5327
Record Dates: First submitted 2019-04-26; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-04

CONDITIONS: Cleft Palate
Keywords: cleft palate; velopharyngeal sphincter; velopharyngeal insufficiency; speech therapy; rehabilitation
MeSH Terms: conditions — Cleft Palate; Velopharyngeal Insufficiency; Communication Disorders

STUDY DESIGN:
Intervention Model Description: Uncompared before-after clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group before-after (Experimental): Speech therapy with Semiocluded vocal tract exercise.
  Interventions: Behavioral: Group before-after

INTERVENTIONS:
Behavioral: Group before-after — The group was submitted to four weeks of speech therapy intervention with Semiocluded vocal tract exercise. The 12 participants were evaluated before and after the intervention with a multidimensional evaluation comprised of analysis of images generated by specialized videonasoendoscopy software, analysis of speech emissions by perceptual-auditory evaluation and acoustic analysis, and vocal self-assessment.

SUMMARY:
Analyze the effect of SOVTE (Semi-occluded Vocal Tract Exercise), with high resistance tube, on the velopharyngeal mechanism, for speech rehabilitation of twelve patients with cleft palate with vocal alterations, after four weeks. The study was developed in the city of Porto Alegre, southern Brazil. The hypothesis of the study is that after four weeks of exclusive therapy with exercise it will be improvement in the voice of patients with cleft palate.

DETAILED DESCRIPTION:
The study is an uncompared before-after clinical trial. All patients were submitted to videonasoendoscopy and had their vocal emissions recorded before and after the four weeks of speech therapy. These individuals were submitted to multidimensional evaluation comprised of analysis of images generated by specialized videonasoendoscopy software, analysis of speech emissions by perceptual-auditory evaluation and acoustic analysis, and vocal self-assessment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with surgically repaired CLP (Cleft lip and palate), regardless of gender and regardless of the type of clef palate.
* The sample only included patients aged 6+ because this is the ideal age to be submitted to videonasoendoscopy.
* These patients attended four speech therapy sessions.
* All individuals agreed to participate in this research voluntarily.

Exclusion Criteria:

* Individuals with cleft lip and palate associated with genetic syndromes or other congenital malformation
* Individuals who proved unable to do SOVTE (Semi-occluded Vocal Tract Exercise),
* No condition to be submitted to videonasoendoscopy examination,
* Patients who did not attend the four sessions of therapy or who did not do exercise at home were excluded from the sample.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Analyze the effect of semi-occluded vocal tract exercise, with high resistance tube, on the velopharyngeal mechanism | one month
  Patients were submitted to evaluation of the VPS (velopharyngeal sphincter) region before and after the speech therapy. Patients were sitting in the examination chair, facing the examiner, throughout the entire procedure. The otorhinolaryngologist framed the image of the VPS and tried to maintain the optic fiber positioned at this site while those being evaluated performed selected sentences.

SECONDARY OUTCOMES:
Changes on speech after semi-occluded vocal tract exercise in cleft palate. | one month
  To measure this outcome, samples of the participant's speech were recorded before and after the exercise with semi-occluded vocal tract (SOVTE). The vocal samples were randomly presented to three experients judges, voice specialists. They analyzed the samples and consensually completed the protocol of perceptual-auditory evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Vinicius M Collares, MD, PhD, Study Director — Chief of plastic surgery of Clinicas Hospital of Porto Alegre's

IPD SHARING:
Plan to Share IPD: No
The IPD was analysed and will be published in conjunction.